CLINICAL TRIAL: NCT00599391
Title: Phase 1 Study to Examine the Use of Far Infrared Radiation for Renal Failure.
Brief Title: Far Infrared Treatment for Kidney Diseases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-RF-CTP1
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Kidney Failure
Keywords: KIDNEY FAILURE, ACUTE; KIDNEY FAILURE, CHRONIC; RENAL INSUFFICIENCY
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Far Infrared Radiation
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared Radiation for 30 to 40 minutes per session.

SUMMARY:
Renal failure or kidney failure is a situation in which the kidneys fail to function adequately. It is divided into acute and chronic forms; either form may be due to a large number of other medical problems.

DETAILED DESCRIPTION:
There are many causes of chronic kidney disease. The most common cause is diabetes mellitus. Acute renal failure is a rapidly progressive loss of renal function, generally characterized by body fluids disturbances and electrolyte derangement.

It is believed that far infrared radiation of the central nervous system, the endocrine system and the kidneys will help in the management of renal failure and a possible cure.

ELIGIBILITY:
Inclusion Criteria:

* People with kidney diseases

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Kidney Function Improvement | 1 year

SECONDARY OUTCOMES:
Causes of Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Chair — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada